CLINICAL TRIAL: NCT05980533
Title: Utility and Feasibility of Prehospital Portable Ultrasound to Predict Heart Failure Readmission Risk
Brief Title: Portable Ultrasound to Predict Heart Failure Readmission Risk
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started and research team member leaving institution
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2307-41
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Patient Readmission
Keywords: Ultrasound
MeSH Terms: conditions — Heart Failure | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Experimental): Ultrasound at hospital discharge and at follow up in 7-10 days
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound at hospital discharge and at follow up at 7-10 days

SUMMARY:
The purpose of this research is to use a handheld ultrasound to assess patients with congestive heart failure (CHF) to see if the ultrasound can help predict readmission to the hospital. The study will include patients who are admitted to the hospital for CHF. Participants will have two ultrasounds at hospital discharge and at a follow up visit.

DETAILED DESCRIPTION:
The purpose of this research is to see if a portable ultrasound can help predict readmission to the hospital for patients who are admitted to the hospital for CHF. The study will enroll patients who take part in Mobile Integrated Healthcare as part of their routine care. Participants will have two ultrasounds. The first ultrasound will be at hospital discharge.

Between seven to ten days after hospital discharge participants will be visited at their home in follow-up as the usual standard of care for Mobile Integrated Healthcare. At this visit participants will have a second ultrasound. Participants will be followed for one year for hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

* Primary admission diagnosis is listed as congestive heart failure, with an acute component of decompensation.
* Age greater than 18 years.
* Principal residence within the geographic reach of our MIH program.

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission | 30 days
  Hospital readmission within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Dewar, Principal Investigator — The Guthrie Clinic

IPD SHARING:
Plan to Share IPD: No